CLINICAL TRIAL: NCT06620185
Title: A Two-arm, Non-randomised, Open-label Experimental Medicine Study to Compare Immune Responses Between Healthy Volunteers Aged 18-40years Receiving Either an Intranasal Live-attenuated Influenza Vaccine or Viral Challenge With GMP Influenza A/Belgium/4217/2015 (H3N2)
Brief Title: GEneRating Mucosal Immunity After INfluenzA Infection and Vaccination in Lung and Lymphoid TissuE
Acronym: GERMINATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23HH8514
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Influenza
Keywords: LAIV; Challenge; Vaccine; Influenza; Flu
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAIV (Experimental)
  Interventions: Biological: FLUENZ
- IAV Challenge (Experimental)
  Interventions: Biological: Influenza challenge virus

INTERVENTIONS:
Biological: FLUENZ — LAIV (Intranasal Influenza Vaccine)
  Other Names: Influenza vaccine; LAIV
  Arms: LAIV
Biological: Influenza challenge virus — Influenza challenge virus (H3N2 strain)
  Arms: IAV Challenge

SUMMARY:
This experimental medicine study aims to compare immune responses in healthy adult volunteers aged 18-40 years against influenza vaccination and infection in the upper and lower respiratory tract, following administration of a live-attenuated influenza vaccine delivered by nasal spray versus influenza A (H3N2) viral challenge.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18-40 years inclusive
* Sero-suitable as defined by a serum micro-neutralisation titre <1:20
* Female participant who is not of child-bearing potential as assessed by an investigator OR is willing and able to use contraception as described in the protocol
* Male participants who are willing to use one of the contraception methods described in the protocol
* In good health with no clinically significant medical conditions

Exclusion Criteria

* History of clinically significant/currently active conditions;

  * Cardiovascular, thromboembolic/cerebrovascular disease.
  * Types of chronic respiratory disease in adulthood.
  * Significant wheeze in the past
  * Respiratory symptoms including wheeze, resulting in hospitalisation
  * Known bronchial hyperactivity to viruses
  * Diabetes mellitus
  * Migraine with associated symptoms like hemiplegia/vision loss. Cluster headache/migraine/prophylactic treatment for migraine.
  * History of autoimmune disease/known immunodeficiency of any cause
  * Immunosuppression.
  * Known coagulation disorder/anticoagulant therapy
  * Psychiatric illness including participants with a history of depression and/or anxiety with associated psychiatric comorbidities
  * Other major disease that, under the PI's discretion, could interfere with the participant completing the study.
* Concurrent serious illness including history of malignancy that could interfere with the study or a participant completing the study.
* Known IgA deficiency/immotile cilia syndrome/Kartagener's syndrome
* Significant abnormality altering the anatomy/function of the nose or nasopharynx, a clinically significant history of epistaxis within the last 3 months, nasal/sinus surgery within 6 months of Day 0, including nasopharyngeal malignancy, arterio-venous malformation, or undiagnosed nasopharyngeal mass
* Inhaled bronchodilator/inhaled steroid use within the last 12 months before Day 0
* Acute upper respiratory tract infection in the past 6 weeks.
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months before Day 0
* Receipt of any vaccine within 30 days of Day -14
* Any significant medical condition/prescribed drug, under the PI's discretion
* Presence of cold-like symptoms and/or fever on Day -14 or Day 0.
* Receipt of blood/blood products/loss (including blood donations) of 550 mL or more of blood during the 3 months prior to Day -14.
* Significant history/presence of drug/alcohol misuse by self-report.
* Current use of drugs through nose inhalation or inhaled route including recreational drugs.
* Regular smoking and/or vaping and/or using nicotine-containing products in the past 3 months OR >5 pack-year lifetime history by self-report (5 pack years is equivalent to one pack of 20 cigarettes per day for 5 years).
* History of anaphylaxis and/or a history of severe allergic reaction or significant intolerance to any food/drug, as assessed by the PI.
* Clinically active rhinitis (including hay fever)/history of moderate to severe rhinitis/history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of enrolment.
* Anyone with any of the following contraindications to receiving the Fluenz Tetra Vaccine:

  * Allergy to gentamicin, gelatin or the other ingredients of the fluenz vaccine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Peak symptoms related to inoculation with a GMP-adherent influenza A (H3N2) virus in healthy adults aged 18-40 | 14 days
  Peak self-reported symptom scores by modified Jackson score from the viral challenge (Day 0) up to Day 14 follow-up
Average duration of symptoms related to inoculation with a GMP-adherent influenza A (H3N2) virus in healthy adults aged 18-40 | 14 days
  Average duration of self-reported symptom scores by modified Jackson score from the viral challenge (Day 0) up to Day 14 follow-up
To confirm symptoms related to inoculation with a GMP-adherent influenza A (H3N2) virus in healthy adults aged 18-40 by Area Under the Curve | 14 days
  Self-reported symptom scores by modified Jackson score from the viral challenge (Day 0) up to Day 14 follow-up (Area Under the Curve)
Peak symptoms related to inoculation with LAIV in healthy adults aged 18-40 | 14 days
  Peak self-reported symptom scores by modified Jackson score from the vaccination (Day 0) up to Day 14 follow-up
Average duration of symptoms related to inoculation with LAIV in healthy adults aged 18-40 | 14 days
  Average duration of self-reported symptom scores by modified Jackson score from the vaccination (Day 0) up to Day 14 follow-up (Peak, Duration, Area Under the Curve)
To confirm symptoms related to inoculation with LAIV in healthy adults aged 18-40 by Area Under the Curve | 14 days
  Delf-reported symptom scores by modified Jackson score from the vaccination (Day 0) up to Day 14 follow-up (Area Under the Curve)

SECONDARY OUTCOMES:
To assess influenza viral dynamics in upper respiratory samples | 28 days
  To assess influenza viral dynamics in upper respiratory samples using Viral load by RT-PCR
To assess antibody levels in blood before and after influenza challenge infection | 28 days
  Antibody levels by ELISA, haemagglutination inhibition assay or microneutralisation
To assess LAIV viral dynamics by RT-PCR in upper respiratory samples | 28 days
  To assess LAIV viral dynamics by RT-PCR in upper respiratory samples using Viral load by RT-PCR
To assess antibody levels in blood before and after LAIV | 28 days
  Antibody levels by ELISA, haemagglutination inhibition assay or microneutralisation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, Imperial College Healthcare NHS Trust, London, United Kingdom